CLINICAL TRIAL: NCT04253535
Title: A Prospective Study to Evaluate the Risk of Recurrence of Cervical Artery Dissection During Subsequent Pregnancies
Brief Title: Risk of Recurrence of Cervical Artery Dissection During Pregnancy and Puerperium
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0267
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Cervical Artery Dissection
Keywords: Pregnancy; Puerperium Recurrence; Cervical artery dissection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaries — Study on questionnaries

SUMMARY:
Cervical artery dissection (CAD) accounts for about 2% of all strokes, and is a major cause of stroke in young people (about 15%). Many cases of CAD during pregnancy and puerperium have been described, suggesting that pregnancy and puerperium may be potential risk factors for CAD. The purpose of this study is to determine whether pregnancy and puerperium are also recurrence risk factors for CAD.

DETAILED DESCRIPTION:
In this study, all women of childbearing age who had had a CAD between 2005 and 2017 are selected. Women are identified using the ICD10 diagnostic coding system. In addition, a text search with key words ("cervical or carotid or vertebral dissection") has been created in a data warehouse of the University Hospital of Nantes.

To determine the recurrence of CAD during pregnancy and puerperium, the participating women will be asked to answer to a questionnaire, by phone or mail. The questionnaire will be conducted by the same investigator, an experienced neurologist. Information about recurrence of CAD, number of pregnancies before and after the event will be recorded, as well as, the site of obstetrical monitoring, way of delivery, and management of antithrombotics, in case of further pregnancy. In case of no further pregnancy after the dissection, the reason will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Extracranial carotid or vertebral dissection
* Symptomatic dissection (with symptom onset within the last four weeks)
* Spontaneous dissection
* Imaging evidence of dissection on MRI/MRA, CTA or ultrasound.

Exclusion Criteria:

* Minors or adults under guardianship
* Intracranial artery dissection
* Traumatic or iatrogenic dissection
* Patient refusal to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Inclusion Criteria:
  * Extracranial carotid or vertebral dissection
  * Symptomatic dissection (with symptom onset within the last four weeks)
  * Spontaneous dissection
  * Imaging evidence of dissection on MRI/MRA, CTA or ultrasound.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Recurrence of CAD during pregnancy, childbirth or puerperium | Day 0
  This primary study endpoint will be evaluated by a questionnaire asked directly to participating women.

SECONDARY OUTCOMES:
To determine the absolute risk of recurrence of CAD in this population. | Day 0
  This secondary endpoint will be evaluated by a questionnaire asked directly to participating women.
To assess obstetrical monitoring, way of delivery, and management of antithrombotics during further pregnancy. | Day 0
  This secondary endpoint will be evaluated by a questionnaire asked directly to participating women.
To study the reasons of absence of pregnancy after a history of CAD | Day 0
  This secondary endpoint will be evaluated by a questionnaire asked directly to participating women.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France